CLINICAL TRIAL: NCT02150005
Title: Effects of Non-surgical Periodontal Treatment on Hemogram, Lipid and Glycemic Profiles of Patients With an Indication for Surgical Coronary Revascularization
Brief Title: Non-surgical Periodontal Treatment on Hemogram, Lipid and Glycemic Profiles in Patients With Coronariopathies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Veiga de Almeida (Other)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government)
Responsible Party: Principal Investigator, Walmir Júnio de Pinho Reis Rodrigues, Researcher, Rio de Janeiro State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UVA71/06
Record Dates: First submitted 2014-05-18; First posted 2014-05-29 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Periodontitis; Coronariopathy
Keywords: periodontal diseases; cardiovascular diseases; periodontitis treatment
MeSH Terms: conditions — Periodontitis; Periodontal Diseases; Cardiovascular Diseases | interventions — Periodontal Index

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Periodontal treatment (Experimental): The test group received oral hygiene instructions, supragingival and subgingival scaling and root planning using curettes and an ultrasonic appliance.
  Interventions: Procedure: Periodontal treatment
- Control (No Intervention)

INTERVENTIONS:
Procedure: Periodontal treatment
  Arms: Periodontal treatment

SUMMARY:
Objective: The aim of this study was to examine the effects of non-surgical periodontal treatment on the hemogram, glycemic and lipid profiles in cardiopathic patients with an indication for surgical revascularization.

Materials and Methods: Twenty-two patients with chronic periodontitis, over 35 years of age (mean age 59.45 years) randomly assigned into 2 groups were evaluated. Test group (n=11), received periodontal treatment before the surgical procedure, and control group (n=11), did not received periodontal treatment prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing cardiovascular treatment;
* Eight viable teeth in the oral cavity;
* Four periodontal sites with periodontal probing depths ≥5mm in different teeth.

Exclusion Criteria:

-

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Reduction in probing depth in sites with PPD>3mm | Baseline and 90 days after the initial exam
  Reduction of 11.4% in probing depth in sites with Periodontal Probing Depth>3mm
Reduction in probing depth in sites with PPD>5mm | Baseline and 90 days after the initial exam
  Reduction of 6.3% in probing depth in sites with Periodontal Probing Depth>5mm
Reduction in probing depth in sites with CAL>3mm | Baseline and 90 days after the initial exam
  Reduction of 4.6% in probing depth in sites with Clinical Attachment Level >3mm.
Reduction in probing depth in sites with CAL >5mm | Baseline and 90 days after the initial exam
  Reduction of 3.6% in probing depth in sites with Clinical Attachment Level >5mm.
Leukocyte count | Baseline and 90 days after the initial exam
  Non-significant reduction of leukocyte count in the test group. Mean difference of 74.6 m/mcL.
Glucose | Baseline and 90 days after the initial exam
  Glucose showed a non-significant increase in the test group. Mean difference of 24.2 mg/dL.
Hemocyte | Baseline and 90 days after initial exam
  Hemocyte presented a non-significant reduction in the test group. Mean difference 0.39 m/mcL
Hemoglobin | Baseline and 90 days after initial exam
  Non-significant reduction in test group. Mean difference of 0.2 g/dL
Total Cholesterol | Baseline and 90 days after initial exam
  Significant reduction in the test group. Mean reduction of 27.4 mg/dL.
High density lipid | Baseline and 90 days after initial exam
  Significant reduction in test group. Mean difference of 8.2 mg/dL.
Low density lipid | Baseline and 90 days after initial exam
  Non-significant reduction in test group. Mean difference of 8.9 mg/dL.